CLINICAL TRIAL: NCT06938763
Title: A Phase I, Randomized, Double-blinded, Placebo-Controlled First-in-human Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of J4 Dry Powder Capsule After Oral Administration of Single and Multiple Ascending Doses to Healthy Adults
Brief Title: Evaluation of the Safety, Tolerability, and Pharmacokinetics of J4 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NRT001-P1-001-2024
Record Dates: First submitted 2025-03-06; First posted 2025-04-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimers; Disease; Disorder
MeSH Terms: conditions — Alzheimer Disease; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- J4 Cohort 1 (Experimental)
  Interventions: Drug: J4
- J4 Cohort 2 (Experimental)
  Interventions: Drug: J4
- J4 Cohort 3 (Experimental)
  Interventions: Drug: J4
- J4 Cohort 4 (Experimental)
  Interventions: Drug: J4
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: J4 — dry powder capsule
  Arms: J4 Cohort 1; J4 Cohort 2; J4 Cohort 3; J4 Cohort 4
Drug: Placebo — Placebo dry powder capsule
  Arms: Placebo

SUMMARY:
A Phase I, Randomized, Double-blinded, Placebo-Controlled First-in-human Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of J4 Dry Powder Capsule after Oral Administration of Single and Multiple Ascending Doses to Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between 18 and 64 (inclusive) years of age at the time of consent
2. Body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive); male subjects must weigh a minimum of 50 kg while female subjects must weigh a minimum of 45 kg.
3. Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, vital sign measurement, ECG, and clinical laboratory test results.
4. Male subjects with a female partner of childbearing potential are eligible to participate if they meet either of the following conditions:

   * They are surgically or biologically sterile (surgically sterile is defined as vasectomy with documented negative semen analysis/azoospermia).
   * They commit to the use of highly effective methods of contraception (defined as those that, alone or in combination, result in a failure rate less than 1 percent per year) from study Day -1 until 90 days after the last dose of the study drug. Male subject must use a condom, and the subject's female partner must use either an occlusive cap (cervical cap or diaphragm) with spermicide or an intrauterine device.
   * They are abstinent from intercourse from study Day -1 until 90 days after the last dose of the study drug.
5. Male subjects must agree to refrain from sperm donation and females refrain from ova donation from Study Day -1 until 90 days after the last dose of the study drug.
6. Female subjects of childbearing potential (which is defined as any woman or adolescent who has begun menstruation) are eligible to participate if they meet either of the following conditions:

   * They are surgically of biologically sterile (surgically sterile is defined as the subject has one of the following: documented hysterectomy, documented bilateral salpingectomy, documented bilateral oophorectomy). If they have undergone tubal ligation, the procedure must have occurred at least 6 weeks prior to the 1st study drug administration.
   * They commit to use of highly effective methods of contraception, starting from at least 30 days prior to 1st study drug administration and continuing for at least 90 days after the last dose of the study drug. The highly effective methods include the use of condom by the male partner, in combination with one of the following by the female participant:

     * Occlusive cap (cervical cap or diaphragm) with spermicide
     * Intrauterine device
   * The subject has a vasectomized male partner with documented negative semen analysis/azoospermia, provided that the partner is the sole sexual partner of the female subject.
   * They perform sexual abstinence from at least 30 days prior to the 1st study drug administration and until at least 90 days after the last dose of the study drug.
7. Female subjects of postmenopausal state must be amenorrhea for at least 2 years or have no menses for 12 month and a high FSH level in postmenopausal range.
8. Provide signed informed consent prior to any study procedures commencing, understand and comply with the requirements of the study, and be able to communicate with the investigator.

Exclusion Criteria:

Subject with any of the following will be excluded from the study.

1. Female who are pregnant or breastfeeding or have a positive pregnancy test at screening, admission or prior to study drug administration.
2. A history of any significant medical illness, including but not limited to neurological, cardiovascular, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic, or renal disease; a history of cancer within the past 5 years.
3. Any clinically significant ECG abnormalities at screening (e.g., QTcFd > 440 ms in men or QTcFd > 460 ms in women).
4. Subjects with blood pressure outside the normal range of 90-140 mm Hg for systolic or 50-90 mm Hg for diastolic at screening.
5. Subjects with a history of cardiovascular disease, such as arrhythmia, hypertension, hypotension, angina pectoris, myocardial infarction, or heart failure.
6. Any lab values that suggest clinically significant hepatic abnormalities (ALT, AST, or TBL ≥ 1.1 ULN) or renal dysfunction (Cr ≥ 1.5 mg/dL) at screening.
7. Clinically significant acute illness or infection within 14 days prior to Day -1.
8. Current or recent (within 3 months) gastrointestinal disease, including gastrointestinal ulceration, gastroesophageal reflux disease, gastritis, or any gastrointestinal surgery that could impact the absorption of the study drug.
9. Any major surgery within 4 weeks prior to 1st study drug administration
10. Blood donation of approximately 250 ml or more within 8 weeks prior to study drug administration, or 500 ml or more within 12 weeks prior to study drug administration, or plasma donation within 2 weeks prior to study drug administration.
11. Inability to tolerate oral medication.
12. Inability to be venipunctured and/or tolerate venous access.
13. Subjects has had any use of tobacco- or nicotine-containing products within 6 months prior to screening.
14. Subjects with daily caffeine intake of more than 200 mg/day (about 2 cups of coffee, 1 cup equals to 8 ounces or about 240 mL) over the past 6 months.
15. Subjects with alcohol consumption of > 1 drink daily over the past 6 months. One drink of alcohol is found in 12 ounces (355 mL) of regular beer (about 5% alcohol), 5 ounces (148 mL) of table wine (about 12% alcohol), and 1.5 ounces (44 mL) of distilled spirits (about 40% alcohol).
16. Recent (within 6 months) drug or alcohol abuse
17. History of any significant drug allergy
18. Positive blood screen for HCV, HBV or HIV
19. Positive urine screen for drugs of abuse or alcohol serum test
20. Exposure to any investigational drug within 4 weeks prior to study drug administration
21. Use of any prescription drugs and other drugs, including over-the-counter medications, herbal preparations, and dietary supplements within 2 weeks or 5 half-lives of the drug, whichever is longer, prior to study drug administration.
22. Receipt of any protein- or antibody-based therapeutic agents (e.g., growth hormones or monoclonal antibodies) within 3 months before study drug administration. People who have received flu or SARS-CoV-2 vaccination within 4 weeks prior to the 1st study drug administration.
23. Use of an oral, injectable or implantable hormonal contraceptive agent within 14 days prior to study drug administration.
24. (MAD only) "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

    * Suicidal Ideation Item 3 (active suicidal ideation with any methods [not plan] without intent to act)
    * Suicidal Ideation Item 4 (active suicidal ideation with some intent to act, without specific plan)
    * Suicidal Ideation Item 5 (active suicidal ideation with specific plan and intent)
    * Any of the Suicidal Behavior items (actual attempt, interrupted attempt, aborted attempt, preparatory acts or behavior) "Yes" responses for any of the following items on the C-SSRS (within past 12 months):
    * Suicidal Ideation Item 1 (wish to be dead)
    * Suicidal Ideation Item 2 (non-specific active suicidal thoughts) Serious risk of suicide in the opinion of the investigator is also exclusionary.
25. Any reason or opinion of the investigator that would prevent the subject from participation in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Day 1 to Day 14
  Vital signs, 12-lead ECGs, clinical laboratory testing, and adverse events (C-SSRS evaluation for MAD only) will be assessed.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5; (MAD) Day 1 to Day 8
  maximum concentration (Cmax)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5; (MAD) Day 1 to Day 8
  time to maximum concentration (Tmax)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5; (MAD) Day 1 to Day 8
  AUC from time 0 to 24 hours post-dose (AUC0-24)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5; (MAD) Day 1 to Day 8
  half-life (T1/2)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5; (MAD) Day 1 to Day 8
  mean residence time (MRT)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5; (MAD) Day 1 to Day 8
  area under the concentration-time curve (AUC) from time 0 to infinity (AUC0-∞)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5
  AUC from time 0 to last quantifiable concentration (AUC0-last)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5
  Apparent clearance (CL/F)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (SAD) Day 1 to Day 5
  apparent volume of distribution (Vd/F)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (MAD) Day 1 to Day 8
  maximum concentration (Cmax) concentration at the end of dosing interval (Ctrough)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (MAD) Day 1 to Day 8
  AUC over the dosing interval (AUC0-τ)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (MAD) Day 1 to Day 8
  apparent clearance at the steady state (CLss/F)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (MAD) Day 1 to Day 8
  apparent volume of distribution (Vd/F)
Pharmacokinetics (PK) of J4 Dry Powder Capsule | (MAD) Day 1 to Day 8
  accumulation ratio (Racc)

OTHER OUTCOMES:
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  maximum concentration (Cmax)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  time to maximum concentration (Tmax)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  area under the concentration-time curve (AUC) from time 0 to infinity (AUC0-∞)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  AUC from time 0 to 24 hours post-dose(AUC0-24)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  AUC from time 0 to last quantifiable concentration (AUC0-last)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  Apparent clearance (CL/F)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  apparent volume of distribution (Vd/F)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  half-life (T1/2)
Effect of food on J4 Dry Powder Capsule bioavailability | Day 1 to Day 10
  mean residence time (MRT)

CONTACTS AND LOCATIONS:
Overall Officials: Yijuang Chern, Director of Institute of Biomedical Sciences, PhD, Study Director — Academia Sinica, Taiwan
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No